CLINICAL TRIAL: NCT05036317
Title: Empagliflozin for the Treatment of Postprandial Hypoglycemia
Acronym: EmpHy
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Early terminated after prespecified interim analysis due to lack of efficacy. No relevant safety signals.
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021-00078; kt21Donath
Record Dates: First submitted 2021-09-01; First posted 2021-09-05 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Postprandial Hypoglycemia
Keywords: Empagliflozin; bariatric surgery; hyperinsulinemic response; SGLT2-inhibitor; insulin secretion; postbariatric hypoglycemia
MeSH Terms: conditions — Hypoglycemia | interventions — empagliflozin

STUDY DESIGN:
Intervention Model Description: 1:1 randomized, placebo-controlled, parallel-group double-blind superiority trial
Who Masked: Participant, Investigator
Masking Description: Both subjects and investigators will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Empagliflozin (Experimental): Standard dose of empagliflozin (Jardiance®; Boehringer Ingelheim GmbH), i. e. 10 mg. Empagliflozin is an orally available inhibitor of SGLT2 and approved for the treatment of type 2 diabetes mellitus and will be given per os once daily in the morning for 28 days.
  Interventions: Drug: Empagliflozin (Jardiance®;
- Placebo (Placebo Comparator): Placebo provided by Boehringer Ingelheim Switzerland. Per os once daily in the morning for 28 days.
  Interventions: Other: Placebo Control Intervention

INTERVENTIONS:
Drug: Empagliflozin (Jardiance®; — Each tablet contains the active substance of 10 mg empagliflozin as well as the adjuvant lactose-monohydrate and is taken orally once daily in the morning.
  Arms: Empagliflozin
Other: Placebo Control Intervention — Placebo will be provided by Boehringer Ingelheim. It is identical to the interventional product apart from the active compound.
  Arms: Placebo

SUMMARY:
This randomized trial is to test whether a treatment with empagliflozin is superior to placebo in patients with postprandial hypoglycemia after bariatric surgery, that is if it improves health related quality of life (mentally or physically) or reduces the risk of hypoglycemic events.

DETAILED DESCRIPTION:
Postprandial hypoglycemia is a debilitating medical complication after bariatric surgery for which no approved pharmacological treatment exists. The prevalence of hypoglycemia in bariatric patients ranges from 0.5 % severe episodes up to 56 % and its symptoms range from asymptomatic to deleterious. This hypoglycemic condition is characterized by a rapid increase of plasma glucose after carbohydrate ingestion followed by an exaggerated hyperinsulinemic response. Hypoglycemia itself may lead to increased hunger, carbohydrate ingestion and following weight regain.

In a placebo-controlled, randomized, double-blind, crossover study, the SGLT2-inhibitor empagliflozin statistically significantly reduced the number of symptomatic hypoglycemia (2 vs. 7 symptomatic hypoglycemic episodes; p=0.013) compared to placebo after a mixed meal test in 12 patients after Roux-en-Y gastric bypass. Empagliflozin reduced the postprandial rise in glycemia and decreased subsequent insulin secretion, underlining the postulated mechanism of action.

This randomized trial is to test whether a treatment with empagliflozin is superior to placebo in patients with postprandial hypoglycemia after bariatric surgery, that is if it improves health related quality of life (mentally or physically) or reduces the risk of hypoglycemic events.

ELIGIBILITY:
Inclusion Criteria:

* Patients after bariatric surgery (i.e. sleeve gastrectomy, Roux-en-Y gastric bypass, omega- loop bypass, biliopancreatic diversion) with documented hypoglycemia, i. e. < 3.0 mmol/l and at least 5 hypoglycemic episodes per week despite dietary modification
* For women with child-bearing potential, willingness to use contraceptive measures adequate to prevent pregnancy during the study
* Informed Consent as documented by signature

Exclusion Criteria:

* Any type of diabetes mellitus according to ADA criteria
* Intolerance to the study drug
* Signs of current infection
* Use of any drug therapy for postbariatric hypoglycemia apart from acarbose (all remaining drugs have to be discontinued four half-life times before screening phase)
* Neutropenia (leukocyte count < 1.5 × 109/L or absolute neutrophil count (ANC) < 0.5 × 109/L)
* Anemia (hemoglobin < 11 g/dL for males, < 10 g/dL for females)
* Clinically significant kidney or liver disease (creatinine > 1.5 mg/dL, AST/ALT > 2 × ULN, alkaline phosphatase > 2 × ULN, or total bilirubin [tBili] > 1.5 × ULN)
* Uncontrolled congestive heart failure
* Uncontrolled malignant disease
* Currently pregnant or breastfeeding
* Known or suspected non-compliance, drug or alcohol abuse
* Meeting the criteria for vulnerability (e.g. participants incapable of judgment or participants under tutelage)
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc.
* Participation in another clinical trial using investigational drugs in the last 30 days or planned participation in the next 60 days
* Previous enrolment into the current study,
* Enrolment of the investigator, his/her family members, employees and other dependent persons

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-03-11 (Actual); Primary Completion 2024-08-05 (Actual); Study Completion 2024-08-05 (Actual)

PRIMARY OUTCOMES:
Change in Quality of life (mental health; as assessed by the SF-36 mental health component score; MCS) | at baseline, at day 29 and at day 60 (+/- 10 days) after baseline
  Change in Quality of life (mental health; as assessed by the SF-36 mental health component. Each item is scored on a 0 to 100 range so that the lowest and highest possible scores are 0 and 100, respectively. Scores represent the percentage of total possible score achieved.
Change in Quality of life (physical health; as assessed by the SF-36 mental physical component score; PCS) | at baseline, at day 29 and at day 60 (+/- 10 days) after baseline
  Change in Quality of life (physical health; as assessed by the SF-36 mental physical component score; PCS). Each item is scored on a 0 to 100 range so that the lowest and highest possible scores are 0 and 100, respectively. Scores represent the percentage of total possible score achieved.
Hypoglycemic events defined as glucose values below 3.0 mmol/l | at 28 days after randomization
  Hypoglycemic events defined as glucose values below 3.0 mmol/l

SECONDARY OUTCOMES:
Postprandial Symptoms of hypoglycemia defined as acute onset of typical symptoms according to Edinburgh Hypoglycemia Scale along with a decreasing blood glucose level. | at 28 days after randomization
  Postprandial Symptoms of hypoglycemia defined as acute onset of typical symptoms according to Edinburgh Hypoglycemia Scale (7-point Likert scale (1 = not present, 7 = very intense)) along with a decreasing blood glucose level. The postprandial period is defined as 3 hours following meal intake.
Hypoglycemia unawareness (measured by modified Clarke Score) | at 28 days after randomization
  Hypoglycemia unawareness (measured by modified Clarke Score). The Clarke method comprises eight questions characterizing the participant's exposure to episodes of moderate and severe hypoglycemia. It also examines the glycemic threshold for, and symptomatic responses to, hypoglycemia. A score of four or more implies impaired awareness of hypoglycemia.
Fear of hypoglycemia (measured on a scale of 0 to 10) | at 28 days after randomization
  Fear of hypoglycemia (measured on a scale of 0 to 10)
Time below range (TBR): % of sensor glucose readings and time between 3.0 and 3.8 mmol/L) | at 28 days after randomization
  Time below range (TBR): % of sensor glucose readings and time between 3.0 and 3.8 mmol/L)
Time in hypoglycemia: % of sensor glucose readings and time below 3.0 mmol/L | at 28 days after randomization
  Time in hypoglycemia: % of sensor glucose readings and time below 3.0 mmol/L
Pattern of sensor glucose | at 28 days after randomization
  Pattern of sensor glucose, defined as the slope of postprandial increase (calculated as the maximal rate of increase observed over 20min in the postprandial period) and decrease (calculated as the maximal rate of decrease over 20min in the postprandial period).
Glycemic variability | at 28 days after randomization
  Glycemic variability (defined as the coefficient of variation (CV) of sensor glucose)
Mean amplitude of sensor glucose excursions (MAGE) | at 28 days after randomization
  Mean amplitude of sensor glucose excursions (MAGE)
Total number of adverse events | up to 60 days after randomization
  Total number of adverse events
Number of Serious adverse events | up to 60 days after randomization
  Number of Serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Marc Y Donath, Prof. Dr. med., Principal Investigator — University Hospital Basel, Division of Endocrinology, Diabetes and Metabolism
Locations (3):
- Switzerland (3):
  - University Hospital Basel, Division of Endocrinology, Diabetes and Metabolism, Basel
  - University Hospital Berne and Center of Bariatric Surgery Berne, Bern
  - Cantonal Hospital Olten, Endocrine Outpatient Clinic, Olten